CLINICAL TRIAL: NCT05532163
Title: A Prospective, Multicenter, Interventional, Open-Label, Single-arm Phase IV Study Over 24 Weeks to Investigate the Radiological Onset of Action After Treatment Initiation With Subcutaneous Natalizumab in Patients With Relapsing-Remitting Multiple Sclerosis (TYS-ON)
Brief Title: A Study to Investigate the Radiological Onset of Action After Treatment Initiation With Subcutaneous (SC) Natalizumab in Participants With Relapsing-Remitting Multiple Sclerosis (RRMS)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DE-TYS-12072; 2022-001820-14 (EudraCT Number)
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Natalizumab (Experimental): Participants will receive natalizumab 300 milligrams (mg) (2*150 mg), SC injection, once every 4 weeks (Q4W) up to Week 24.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Administered as specified in the treatment arm
  Other Names: Tysabri; BG00002

SUMMARY:
The primary objective of this study is to evaluate the radiological efficacy of SC natalizumab over time through Week 24 in natalizumab-naïve participants, as measured by brain magnetic resonance imaging (MRI). The secondary objectives of this study are to evaluate additional lesion-related radiological efficacy measures over time, relapse-based clinical efficacy measures, disability improvement and worsening (EDSS), pharmacokinetic and pharmacodynamic parameters, the immunogenicity of repeated doses, and safety in treatment-naïve participants of SC natalizumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of RRMS according to the McDonald criteria
* Treatment-naïve in respect to natalizumab as disease modifying monotherapy for RRMS
* No or not more than one prior MS disease-modifying therapy
* Highly active RRMS, as defined by at least one relapse in the previous year and at least one T1 gadolinium-enhancing lesion or ≥3 new or enlarging T2 lesions
* EDSS score ≤ 5.5 at Screening
* Estimated glomerular filtration rate (eGFR) >30 millilitre per min (mL/min), as estimated using the Cockcroft-Gault formula.

Key Exclusion Criteria:

* Primary- and secondary-progressive MS
* Participants for whom MRI is contraindicated
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic (including diabetes), urologic, pulmonary, neurologic (except for RRMS), dermatologic, psychiatric, renal, or other major disease that would preclude participation in a clinical study
* History of severe allergic or anaphylactic reactions or known hypersensitivity to any antibody drug therapy.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Cumulative Number of Active Lesions (CUALs) Through Week 24 | Up to Week 24
  Cumulative number of active lesions will be calculated as the sum of the number of gadolinium (Gd)-enhancing lesions and new or enlarging T2 hyperintense lesions that are non-enhancing on post-gadolinium T1-weighted (T1w) scans. It is also referred to as combined unique active lesions (CUALs).

SECONDARY OUTCOMES:
Cumulative Number of CUALs Through Weeks 4, 8, and 12 | Weeks 4, 8, and 12
  CUALs will be calculated as the sum of the number of Gd-enhancing lesions and new or enlarging T2 hyperintense lesions that are non-enhancing on post-gadolinium T1w scans.
Absolute Number of CUALs at Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
  CUALs will be calculated as the sum of the number of Gd-enhancing lesions and new or enlarging T2 hyperintense lesions that are non-enhancing on post-gadolinium T1w scans.
Mean Change From Baseline of CUALs at Weeks 4, 8, 12, and 24 | Baseline, Weeks 4, 8, 12, and 24
  CUALs will be calculated as the sum of the number of Gd-enhancing lesions and new or enlarging T2 hyperintense lesions that are non-enhancing on post-gadolinium T1w scans.
Cumulative Number of New Gd-Enhancing Lesions Through Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
  Cumulative number will be calculated as the sum of the number of Gd-enhancing lesions through Weeks 4, 8, 12, and 24.
Absolute Number of New Gd-Enhancing Lesions at Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
Absolute Number of Persisting Gd-Enhancing Lesions at Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
Absolute Number of Any (New or Persisting) Gd-Enhancing Lesions at Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
Change From Baseline of Any (New or Persisting) Gd-Enhancing Lesions at Weeks 4, 8, 12, and 24 | Baseline, Weeks 4, 8, 12, and 24
Cumulative Number of New or Enlarging T2 Lesions at Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
  Cumulative number will be calculated as the sum of the number of new or enlarging T2 hyperintense lesions through Weeks 4, 8, 12, and 24.
Absolute Number of New or Enlarging T2 Lesions at Weeks 4, 8, 12, and 24 | Weeks 4, 8, 12, and 24
Change From Baseline of New or Enlarging T2 Lesions at Weeks 4, 8, 12, and 24 | Baseline, Weeks 4, 8, 12, and 24
Annualized Relapse Rate | Week 24
  Multiple sclerosis (MS) relapse is defined as the onset of new or recurrent neurological symptoms lasting at least 24 hours, accompanied by new objective abnormalities on a neurological examination, and not explained solely by non-MS processes such as fever, infection, severe stress, or drug toxicity. ARR is defined as the total number of relapses divided by the total participant-time at risk of relapse.
Time to First Relapse | Up to Week 24
  MS relapse is defined as the onset of new or recurrent neurological symptoms lasting at least 24 hours, accompanied by new objective abnormalities on a neurological examination, and not explained solely by non-MS processes such as fever, infection, severe stress, or drug toxicity. Time to first MS relapse will be calculated as the date from first study drug administration through the date of the first relapse, if applicable.
Number of Participants With Expanded Disability Status Scale (EDSS) Improvement and Stable Disease and Worsening at Weeks 12, and 24 | Baseline, Weeks 12, and 24
  The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS. Stable disease is defined as +/- 0.5 change of EDSS. Worsening is > 0.5 increase of EDSS.
Trough Serum Natalizumab Concentration (Ctrough) | Pre dose on Baseline, Weeks 4, 8, 12, and 24
Trough alpha 4 (α4) Integrin Saturation | Pre dose on Baseline, Weeks 4, 8, 12, and 24
Change From Baseline in Lymphocyte Subsets Count | Baseline up to Week 24
  Lymphocyte subsets include T cells, B cells and natural killer cells (cluster of differentiate 4 [CD4], CD8, CD19, and CD56).
Change From Baseline in Anti-Natalizumab Antibodies | Pre dose on Baseline, Weeks 12, and 24
Persistence of Anti-Natalizumab Antibodies | Re-test after 6 weeks of first positive result (up to Week 24)
  Re-test will be done for antibodies after 6 weeks of first positive result.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 24
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Neurologische Praxis Dr. med. Boris-Alexander Kallmann, Bamberg
  - Neurologische Studiengesellschaft Bonn GbR, Bonn

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/